CLINICAL TRIAL: NCT02368730
Title: Documentation of the Efficacy of Desmopressin (MINIRIN Parenteral 4 Microgram/ml Solution for Injection) Within the Context of Surgical Procedures
Brief Title: Documentation of the Efficacy of Desmopressin Within the Context of Surgical Procedures
Acronym: RAPID
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000149
Record Dates: First submitted 2015-02-16; First posted 2015-02-23 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Platelet Dysfunction
MeSH Terms: interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- desmopressin: Treatment according to standard clinical practice.
  Interventions: Drug: desmopressin

INTERVENTIONS:
Drug: desmopressin
  Other Names: Minirin

SUMMARY:
In this non-interventional multicentre, prospective, observational cohort study, the efficacy of desmopressin is evaluated in patients with platelet dysfunction due to acetylsalicylic acid or cox-1-inhibitors within the context of surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Pre-, peri- or postoperative treatment with a standard dose of desmopressin as a result of platelet dysfunction (disturbance of blood platelet function) due to treatment with acetylsalicylic acid or cox-1-inhibitor.
* Decision on the therapy with MINIRIN parenteral 4 Microgram/ml solution for injection has already been made independently by the physician beforehand
* The patients (≥ 18 years) have been informed about the non-interventional study and have given their written consent for participation

Exclusion Criteria:

* Participation in a clinical trial
* Treatment with acetylsalicylic acid for cardiovascular indications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital doctors specialised in anaesthesia
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in platelet function pre- and post-administration of desmopressin | From baseline up to 7 days
  As measured by Platelet Function Analyzer (PFA) 100/200

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (1):
- Charité - Universitätsmedizin Berlin (there may be other sites in this country), Berlin, Germany